CLINICAL TRIAL: NCT05834153
Title: Comparative Effects of Kinesiotaping and Electrical Muscle Stimulation on Low Back Pain and Disability Associated With Diastasis Recti
Brief Title: Effects of Kinesiotaping and Electrical Muscle Stimulation on Low Back Pain and Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0523
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: kinesiotaping; electrical muscle stimulation; low back pain; diastasis recti; exercises
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotaping (Experimental)
  Interventions: Device: kinesiotaping
- electrical muscle stimulation (Active Comparator)
  Interventions: Device: electrical muscle stimulation

INTERVENTIONS:
Device: kinesiotaping — This group underwent a KT application on rectus abdominis muscle (RAM), oblique abdominal muscles (OAM) and cesarean incision twice a week for a period of 4 weeks. First, the scar technique will apply using I band with a tension of 50 % on cesarean incision when the patient will be in supine position. Then, tape will apply on RAM using muscle technique from origin to insertion of the muscle with a tension between 15 and 25 %.
  Band will start on symphysis pubis with no tension, and then the patient was asked to stretch the abdominal region by deep abdominal respiration, and it will ended on xiphoid process.
  Finally, it will perform on the right and left external oblique muscles. The procedure will start with no tension from the bottom end of the 6-12th ribs and then the hip will placed in flexion and rotation to the opposite direction and the band will taped on pubic bone with a tension between 15 and 25 %
  Arms: kinesiotaping
Device: electrical muscle stimulation — It consists of 24 patients who will receive NMES and core stabilization exercises.
  The subjects will explain to relax their abdominal muscles while application Stimulation will apply by four large rectangular electrodes placed over the origin (pubic crest) and insertion (xiphoid process) of the rectus abdominis muscles bilaterally. Straps will used to fix the electrodes in place. A frequency of 80 pulses/min and with a pulse width of 0.1-0.5ms, will the parameter settings apply in this study. The total time for the application of stimulation will 30mins and until a good enough observable muscle contraction will achieve a gradual increase in intensity will perform
  Arms: electrical muscle stimulation

SUMMARY:
To compare the effects of kinesiotaping and electrical muscle stimulation on low back pain and disability associated with diastasis recti.

ELIGIBILITY:
Inclusion Criteria:

* Diastasis recti more than 2 or 2.5cm
* 6 weeks' postpartum cesarean section females
* Primigravida females
* Low back pain due to DR

Exclusion Criteria:

* Normal vaginal delivery
* Episiotomy
* Multigravida women's
* History of abdominal hernia
* History of any abdominal surgery

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — diastasis recti
Enrollment: 48 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th week
  Numeric pain rating scale (an outcome measure) is a pain screening tool commonly used to assess pain severity using a 0 to 10 scale, with 0 measuring no pain and 10 meaning worst pain
Manual muscle testing MMT | 4th week
  The strength of rectus abdominis muscle will recorded on a 0 to 5-point scale using manual muscle test suggested by Dr. Lovett. The patients will positioned in a supine, crook lying attitude with the arms straight by the side. The subjects will directed to lift and reach upwards till the scapular lower end level and if the subject will able to achieve and hold this position successfully then will ask to perform the next position by crossing the hands over the chest and then leaning forward and lifting the scapula off the table. After the patient achieved this position successfully forward reaching with hands crossed and supporting at the back of the head will perform. The scores will recorded based on the position that the patient could achieve and sustain successfully i.e. scores 3, 4 and 5 respectively for the above mentioned positions
Roland Morris Disability Questionnaire (RMDQ) for disability | 4th week
  The questionnaire was used to measure the level and severity of disability occurring due to low back pain reflected by higher numbers on a 24-point scale. The questionnaire was taken at the beginning and after completion of the protocol and the clinical improvement was calculated based on the score
Caliper method | 4th week
  Inter Recti Distance (IRD): The inter recti distance measurement was done by the use of a skin tone caliper. The IRD was measured at three levels both pre and post protocol, that is 2 or more than 2.5 cm above and below the umbilicus and at the umbilicus

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No